CLINICAL TRIAL: NCT02937142
Title: Cognitive Behavior Group Therapy in Adolescents (14-18 Years) With Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: Cognitive Behavior Group Therapy in Adolescents With Attention Deficit Hyperactivity Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015/2115
Record Dates: First submitted 2016-10-14; First posted 2016-10-18 (Estimated); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: Behavior Therapy; Cognitive Therapy; Adolescents; Psychotherapy, Group
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive behavior group therapy (Experimental): Cognitive behavior group therapy in weekly 1,5 hour sessions during 12 weeks, 8 participants and 2 therapists per group, in addition to education on ADHD, and ADHD medication if indicated.
  Interventions: Behavioral: cognitive behavior group therapy; Other: Treatment as usual
- Controls (Other): Treatment as usual: Education on ADHD, and ADHD medication if indicated.
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: cognitive behavior group therapy — 1,5 hours weekly session during 12 weeks, 8 participants, 2 therapists.
  Arms: Cognitive behavior group therapy
Other: Treatment as usual — Education on ADHD, and ADHD medication if indicated

SUMMARY:
Attention Deficit Hyperactivity Disorder (ADHD) is a neurodevelopmental disorder which starts in childhood and is characterized by symptoms of attention deficit, hyperactivity and impulsivity. Persistence into adolescence is frequently associated with among other low educational achievement, interpersonal difficulties, anxious and depressive symptoms and sleep problems. Treatment guidelines recommend psychological treatment as part of the treatment plan, however compared to children and adults, there is still a substantial lack of knowledge about appropriate psychological treatment in adolescents. The present study examines a psychological intervention for adolescents with ADHD, cognitive behavior group therapy. The intervention consists of 12 weekly cognitive behavioral therapy sessions addressing core difficulties and concerns of the adolescent population with ADHD. The investigators wish to determine the efficacy of group therapy in adolescents with ADHD who receive medical treatment but still have impairing ADHD symptoms.

DETAILED DESCRIPTION:
Change February 1st 2017: Inclusion of patients with mild to moderate behavioral problems in order to achieve enough participants in the study.

Change February 1st 2017: The study primarily recruits patients who are on pharmacological treatment for ADHD. However, for ethical reasons and in order to achieve enough participants, the study will also recruit patients who have not responded to at least two drug trials or have been unable to continue pharmacological treatment because of intolerable side effects.

Change February 1st 2018: The Weiss Functional Impairment Rating Scale, Rosenberg and BRIEF questionnaires will not be collected at the 9-month follow-up due to lack of resources (project assistance).

ELIGIBILITY:
Inclusion Criteria:

* Attention deficit hyperactivity disorder (ICD-10)
* Clinical Global Impression (CGI) >=3
* Informed consent patient
* informed consent parents
* if on medication, dosage is stable since at least 2 months

Exclusion Criteria:

* mental retardation
* behavioral problems
* drug addiction
* psychosis
* suicidal

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
ADHD-Rating Scale (ADHD-RS) | 12 weeks (at baseline and immediately after the last group therapy session)
  interview

SECONDARY OUTCOMES:
ADHD-Rating Scale (ADHD-RS) | 9 months
Clinical Global Impression (CGI) | 12 weeks (at baseline and immediately after the last group therapy session)
Weiss Functional Impairment Rating Scale (WFIRS) | 12 weeks (at baseline and immediately after the last group therapy session)
Weiss Functional Impairment Rating Scale (WFIRS) | 9 months
Children's Global Assessment Scale (CGAS) | 9 months
Anxiety symptoms (SCARED) | 12 weeks (at baseline and immediately after the last group therapy session)
Depressive symptoms (Mood and Feelings Questionnaire (MFQ) Norwegian version "Humøret ditt") | 12 weeks (at baseline and immediately after the last group therapy session)
Sleep problems (Adolescent Sleep Wake Scale | 12 weeks (at baseline and immediately after the last group therapy session)
Self-esteem (Rosenberg Self-Esteem Scale) | 12 weeks (at baseline and immediately after the last group therapy session)
Self-esteem (Rosenberg Self-Esteem Scale) | 9 months
Self-efficacy (General Perceived Self-Efficacy Scale) | 12 weeks (at baseline and immediately after the last group therapy session)
Self-efficacy (General Perceived Self-Efficacy Scale) | 9 months
Executive functioning (Behavior Rating Scale of Executive Functioning, BRIEF) | 12 weeks (at baseline and immediately after the last group therapy session)
Executive functioning (Behavior Rating Scale of Executive Functioning, BRIEF) | 9 months
ASEBA Brief Problem Monitor | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Torunn Stene Nøvik, MD PhD, Principal Investigator — St Olavs Hospital University Hospital Trondheim
Locations (1):
- Barne- og ungdomspsykiatrisk poliklinikk, St Olavs Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Novik TS, Haugan AJ, Lydersen S, Thomsen PH, Young S, Sund AM. Cognitive-behavioural group therapy for adolescents with ADHD: study protocol for a randomised controlled trial. BMJ Open. 2020 Mar 25;10(3):e032839. doi: 10.1136/bmjopen-2019-032839. PMID 32213517
- [Derived] Haugan AJ, Sund AM, Young S, Thomsen PH, Lydersen S, Novik TS. Cognitive behavioural group therapy as addition to psychoeducation and pharmacological treatment for adolescents with ADHD symptoms and related impairments: a randomised controlled trial. BMC Psychiatry. 2022 Jun 2;22(1):375. doi: 10.1186/s12888-022-04019-6. PMID 35655149
- See also: Related Info — http://stolav.no/bup